CLINICAL TRIAL: NCT04734288
Title: LIFEHOUSE: a Lifestyle Intervention and Functional Evaluation- a Health OUtcome SurvEy; Description of the Tent Bucket -Immune Support
Brief Title: LIFEHOUSE: Description of the Tent Bucket -Immune Support
Acronym: LIFEHOUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Collaborators: MetaProteomics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-002
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-04

CONDITIONS: Immune Response
Keywords: Nutritional Supplements; Vitamin (Vit.) D3; hs-CRP; Inflammation; Employee wellness program
MeSH Terms: conditions — Inflammation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A single-arm cohort intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immune response (Experimental): This is a single-arm study. All subjects will be treated equally and will receive the same type and amount of nutritional supplements.
  Interventions: Dietary Supplement: Vit.D3 5000 IU, Immune Active

INTERVENTIONS:
Dietary Supplement: Vit.D3 5000 IU, Immune Active — The subjects will receive monthly (for either 3 or 6 months):
  1. Vit.D3 5000 and Immune Active. The first phase includes 3 months of treatment and the second phase includes 6 months of treatment.
  2. An in-home Vit.D/ hs-CRP test kit and asked to self-administer a blood collection via fingerstick and return the kits for analysis within a few days.
  3. Two online questionnaires each month and asked to fill them out within a few days. It will either be the Medical Outcomes Study (MOS) Short Form (SF)-36 and the Health Status Baseline or Health Status Follow-up Questionnaire.
  Other Names: Test kits- Vit.D and hs-CRP blood measurements; Questionnaires

SUMMARY:
This immune support program will be an extension to the existing LIFEHOUSE program. Essential employees in Gig Harbor, WA; Colonial Heights, VA; Lenexa, KS, and Santa Fe Springs, CA, will be offered complimentary supplementation with commercially available nutritional supplements supportive of immune health for several months. The outcome will be measured via blood parameters and questionnaire responses.

DETAILED DESCRIPTION:
This program, as a component of the LIFEHOUSE program, will consist of data collection during a period of supplementation with commercially available nutritional supplements supportive of immune health. Employees, in Gig Harbor, WA; Colonial Heights, VA; Lenexa, KS, and Santa Fe Springs, CA, will be offered the opportunity to participate.

The nutritional and inflammatory status will be captured via fingerstick biomarkers. Participants will receive in-home testing kits including instructions regarding the applicable fingerstick blood collections. Fingerstick testing will include 25-Hydroxy Vitamin D3 (25-OH D3) and high sensitivity c-reactive protein (hs-CRP) measurements at baseline, 1, and 2 (phase 1), or at baseline 1,2, 3, and 6 months intervals (phase 2).

Participants will also be asked to complete applicable questionnaires (QNs) electronically monthly using standard software programs for questionnaire completion.

This will include the Medical Outcome Study (MOS) Short Form (SF) -36 (baseline and monthly) and Health Status QNs including questions on compliance, wellbeing, lifestyle (exercise, shifts worked, medications and supplements, and diet) (baseline and monthly).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 18-69, inclusive
* Metagenics' employees in Gig Harbor, WA; Colonial Heights, VA; Lenexa, KS, and Santa Fe Springs, CA
* General good health
* Willing to give written informed consent to participate in the study

Exclusion Criteria:

* An allergy to any ingredient in Vit.D3 5000 and/or Immune Active
* A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, psychiatric, immunologic/rheumatological, or oncological/hematologic disease.
* Hyperparathyroidism
* Granulomatous disorders including as sarcoidosis, tuberculosis, leprosy, berylliosis, histoplasmosis, and coccidioidomycosis
* Chronic renal insufficiency
* Nephrolithiasis
* Prior cancer diagnosis
* Known infection with human immunodeficiency virus (HIV), tuberculosis (TB), or Hepatitis B or C.
* Established psychiatric disease including moderate to severe depression, thought disorders and bipolar disorder
* Planned use of nutritional supplements (exclusive of multiple vitamin/mineral supplements and medical foods) containing in total more than 1,000 IU Vitamin D3 and/or 10 mg Zinc
* Use of pharmaceutical nitrates for any indication
* Use of drugs of abuse and recreational drugs/substances (such as but not limited to opioids, cocaine, phencyclidine (PCP), and methamphetamine)
* History of marijuana or cannabinoid abuse within 12 months prior to screening and for the duration of the study.
* History of alcohol abuse or a diagnosis of alcoholism within 12 months prior to screening and for the duration of the study.
* Pregnant or breastfeeding women
* Inability to comply with study and/or follow-up visits.
* Any concurrent condition (including clinically significant abnormalities in medical history, physical examination or laboratory evaluations) which, in the opinion of the Principal Investigator (PI), would preclude safe participation in this study or interfere with compliance.
* Any sound medical, psychiatric, and/or social reason which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The benefit of nutritional supplements (Vit.D3 5000, Immune Active) on the improvement of health. | 12 weeks (Phase 1) or up to 6 months (Phase 2)
  The primary objective is to demonstrate the benefit of specific nutritional supplements, Vit.D3 5000 and Immune Active, as measured by demonstrable improvements in health, specifically a marker of nutritional status (25-hydroxy Vitamin D3 (25-OH D3)) and a marker of immune balance (high sensitivity c-reactive protein (hs-CRP) in a real-world setting.

SECONDARY OUTCOMES:
The benefit of nutritional supplements (Vit.D3 5000, Immune Active) on the improvement of quality of life. | 12 weeks (Phase 1) or up to 6 months (Phase 2)
  The first secondary objective is to demonstrate the benefit of specific nutritional supplements, Vit.D3 5000 and Immune Active, as measured by demonstrable improvements in health, specifically upon quality of life as measured by Rand Medical Outcome Study 36-Item Short Form Survey (MOS SF-36).
The benefit of nutritional supplements (Vit.D3 5000, Immune Active) on the improvement of the absence of infections. | 12 weeks (Phase 1) or up to 6 months (Phase 2)
  The second secondary objective is to demonstrate the benefit of specific nutritional supplements, Vit.D3 5000 and Immune Active, as measured by demonstrable improvements in health, specifically experience-defined events (tally of well days during assessed periods and absence of laboratory-confirmed SARS-CoV-2 and Influenza infections).
The benefit of nutritional supplements (Vit.D3 5000, Immune Active) on the improvement of weight and body composition. | 12 weeks (Phase 1) or up to 6 months (Phase 2)
  The third secondary objective is to demonstrate the benefit of specific nutritional supplements, Vit.D3 5000 and Immune Active, as measured by demonstrable improvements in health, specifically in weight and body composition.

CONTACTS AND LOCATIONS:
Overall Officials: Josesph J Lamb, MD, Principal Investigator — Medical Director
Locations (1):
- Personalized Lifestyle Medicine Center, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No